CLINICAL TRIAL: NCT02025491
Title: Efficacy Study of Liposomal Amphotericin in Disseminated Leishmaniasis
Brief Title: Liposomal Amphotericin in Disseminated Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Responsible Party: Principal Investigator, Paulo Roberto Lima Machado, MD PhD, Hospital Universitário Professor Edgard Santos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLLipoBA001
Record Dates: First submitted 2013-12-26; First posted 2014-01-01 (Estimated); Last update posted 2014-01-01 (Estimated); Status verified 2013-12

CONDITIONS: Disseminated Leishmaniasis
Keywords: Disseminated leishmaniasis; Liposomal Amphotericin B; Leishmania braziliensis
MeSH Terms: interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Liposomal Amphotericin (Experimental): Liposomal Amphotericin by intravenous route, 3 to 5 mg/kg/day, during 7 to 14 days of treatment.
  Interventions: Drug: Liposomal Amphotericin B

INTERVENTIONS:
Drug: Liposomal Amphotericin B — Liposomal Amphotericin B will be administered by intravenous route, 3 to 5 mg/kg/day, during 7 to 14 days of treatment. Complete hemogram, aminotransferases (AST, ALT), blood urea and creatinine will be determined in all patients on days -1, and three times/week up to the end of therapy. Patients will bemonitored for side effects daily. Patients will be followed-up at 1, 2, 3, 4 and 6 months post-therapy. Clinical and laboratory adverse events will be graded according to the Common Toxicity Criteria (CTC) of the National Cancer Institute.
  Other Names: Ambisome

SUMMARY:
Disseminated leishmaniasis (DL) is an emerging and severe form of leishmaniasis, with increasing prevalence in Bahia, Brasil. It is characterized by multiple acneiform, papular and ulcerated lesions localized on the face, chest, abdomen and extremities. The number of lesions ranges from 10 to hundreds, and mucosal disease has been documented in more than 40% of the cases.

DL is a hard to cure disease and therapeutic failure with pentavalent antimony has been documented in up to 70% of the cases caused by L. braziliensis in the endemic area of Corte de Pedra, Bahia. The majority of DL patients need several courses of antimony or the use of high dose of Amphotericin B desoxicolate to cure. Therefore DL patients are exposed to relevant drug toxicity, high morbidity due to a long lasting disease, with an important socio-economic impact. Our hypothesis is that liposomal Amphotericin B has a higher cure rate than historic cure rates of pentavalent antimony in the treatment of disseminated leishmaniasis.

ELIGIBILITY:
Inclusion Criteria:

* a) clinical diagnosis of Disseminated Leishmaniasis according to case definition; b) illness duration of less than three months, c) parasite identification by culture or polymerase chain reaction methods, d) no previous treatment for leishmaniasis.

Exclusion Criteria:

* a) immunodeficiency or antibodies to HIV, b) pregnancy or patients not willing or unable to use contraceptives during and 3 months after the end of therapy c) ALT, AST ≥3x normal reference values, creatinine and BUN ≥1.5x normal reference values, d) any evidence of serious underlying disease (cardiac, renal, hepatic, or pulmonary) including serious infection other than DL.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Definitive cure | 3 months after treatment
  Definitive cure at 3 months after the end of treatment is defined as complete epithelialization of all ulcers and complete disappearance of inflammatory infiltrations from all lesions.

SECONDARY OUTCOMES:
Toxicity | During the 7 to 15 days of treatment
  Evaluation of side effects and laboratory parameters during the 7 to 15 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo RL Machado, MD PhD, Principal Investigator — UFBA
Locations (1):
- HUPES, Salvador, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Machado PR, Rosa ME, Guimaraes LH, Prates FV, Queiroz A, Schriefer A, Carvalho EM. Treatment of Disseminated Leishmaniasis With Liposomal Amphotericin B. Clin Infect Dis. 2015 Sep 15;61(6):945-9. doi: 10.1093/cid/civ416. Epub 2015 Jun 5. PMID 26048961